CLINICAL TRIAL: NCT01470677
Title: A Collagen-Fibrin Patch (Tachosil®) for the Prevention of Symptomatic Lymphoceles After Pelvic Lymphadenectomy in Women With Gynecologic Malignancies: a Randomized Clinical Trial
Brief Title: Tachosil for the Prevention of Symptomatic Lymph Cysts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Dr. med. Clemens Tempfer, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TACH-01
Record Dates: First submitted 2011-07-12; First posted 2011-11-11 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Endometrial Cancer; Cervical Cancer
Keywords: lymph cyst; lymphocele; fibrin; collagen; prevention; cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Lymphocele; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- application of Tachosil fibrin patches (Experimental): A Tachosil® patch of 4.8x4.8cm will be attached to the obturator fossa and a Tachosil® patch of 4.8x4.8cm will be attached to the femoral canal of each side of surgery in the intervention group.
  Interventions: Drug: Tachosil fibrin patch
- Control group (No Intervention): In the control group, no Tachosil® patch will be used. No specific drainage of the retroperitoneum will be performed.

INTERVENTIONS:
Drug: Tachosil fibrin patch — A Tachosil® patch of 4.8x4.8cm will be attached to the obturator fossa and a Tachosil® patch of 4.8x4.8cm will be attached to the femoral canal of each side of surgery in the intervention group. In the control group, no Tachosil® patch will be used. No specific drainage of the retroperitoneum will be performed.
  Other Names: EU registration number: EU/1/04/277/002
  Arms: application of Tachosil fibrin patches

SUMMARY:
This is a randomized trial of 140 women with endometrial or cervical cancer undergoing removal of lymph tissue (lymphadenectomy). The application of 4 tachosil fibrin patches to the pelvic side wall after tissue removal is tested against no such intervention after tissue removal. The primary endpoint is to evaluate the incidence of symptomatic pelvic lymphoceles defined by CTCAE 4.03 grade >2 within 4 weeks after surgery in women undergoing open or laparoscopic pelvic lymphadenectomy for cervical and endometrial cancer with and without the application of Tachosil® during surgery. The study's hypothesis is that the application of tachosil fibrin patches will significantly reduce the rate of symptomatic lymph cysts.

DETAILED DESCRIPTION:
1. Background Women with gynecologic malignancies such as cervical and endometrial cancer routinely undergo pelvic lymphadenectomy based on tumor characteristics assessed prior to or during surgery. Pelvic lymphadenectomy may be performed by open surgery or laparoscopy (1-4). Postoperative complications during and after pelvic lymphadenectomy include local abscess, bleeding, lymphocele, and chronic lymphedema of the lower extremities, which has an incidence of 1 to 2% (2,3). In the present trial, we will focus on pelvic lymphoceles, one of the most common complications of pelvic lymphadenectomy. Simonato et al. described a rate of 19/30 (63%) of sonographically detected lymphoceles in men undergoing pelvic extraperitoneal lymphadenectomy for prostate cancer (4). In this trial, 4/19 men with lymphoceles were symptomatic and required medical interventions. In women with cervical cancer, asymptomatic lymphoceles detected by ultrasound have been noted in up to 11% of women after pelvic lymphadenectomy (1,3,5). In 2% of women, clinical symptoms will require a therapeutic intervention (5).

Tachosil® is a fibrin-collagen coated patch and heas been licensed in 2004 and 2007 in Europe for surgical use in humans to support surgical hemostatic interventions. The efficacy and safety of Tachosil® has been demonstrated in liver resection, pulmonary lobectomy, and kidney tumor resection trials (6-8). In men, but not in women, it has been demonstrated that the application of a collagen-fibrin patch to the lymphadenectomy surgery site may prevent a significant proportion of lymphoceles. In a randomized trial, Simonato et al. found that the pelvic application of two Tachosil® patches to the obturator fossa and the femoral canal was sufficient to significantly reduce the rate of sonographically detected lymphoceles within 4 weeks after surgery from 19/30 to 5/30 cases (p=0.001) as well as the mean drainage volume from 190 to 64 ml. Percutaneous puncture of a symptomatic lymphocele was necessary in 1/30 individuals in the intervention group compared to 4/30 individuals in the control group. (4). In women with gynecologic malignancies a single center randomized controlled trial has found, that Tachosil® seems effective to reduce the rate of lymphoceles after pelvic lymphadenectomy (5). 7/30 (23.3%) women in the treatment group compared to 9/28 (57.7%) women in the control group developed asymptomatic lymphoceles (p<0.05) (5). No significant differences between the two groups were observed in the development of symptomatic lymphoceles or the rate of interventions (5). This may be attributable to the small sample size of this study. As symptomatic lymphoceles are more relevant for the patient, it seems clinically more important to the evaluate the impact of Tachosil® on the rate of symptomatic lymphoceles after pelvic lymphadenectomy.

Symptomatic lymphoceles are defined by the CTCA 4.03 grading system as lymphoceles grade >2. This includes all lymphoceles needing medical intervention. Thus this definition comprises, lymphoceles with the presence of localized pelvic pain, pelvic abscess, fever, and/or leg edema in the presence of a sonographically verified pelvic lymphocele.

In summary, the data available in the literature demonstrate that pelvic lymphocles occur in 11 to 63% of individuals undergoing pelvic lymphadenectomy. Symptomatic lymphoceles seem to occur in about 32% of patients undergoing pelvic lymphadenectomy. Intraoperative application of a collagen-fibrin patch may reduce the number of lymphoceles, mean drainage volume, and the necessity of medical interventions such as percutaneous puncture.

Therefore, we intend to perform a multi center randomized clinical trial assessing the efficacy of a collagen-fibrin patch for preventing symptomatic lymphoceles in women undergoing pelvic lymphadenectomy for gynecologic malignancies, ie cervical and endometrial cancer. We hypothesize that, based on the data of Simonato et al. and Tinelli et al., the application of a collagen-fibrin patch (Tachosil®) will reduce the number of symptomatic pelvic lymphoceles by at least 66%.

Primary outcome variable:

2.1. To evaluate the incidence of symptomatic pelvic lymphoceles defined by CTCAE 4.03 grade >2 within 4 weeks after surgery in women undergoing open or laparoscopic pelvic lymphadenectomy for cervical and endometrial cancer with and without the application of Tachosil® during surgery.

Secondary outcome variables:

2.2. To evaluate the incidence of sonographically detected pelvic lymphoceles of at least 2cm in the largest diameter 4 weeks after surgery in women undergoing open or laparoscopic pelvic lymphadenectomy for cervical and endometrial cancer with and without the application of Tachosil® during surgery.

2.3. To evaluate the rate and type of medical interventions for clinically symptomatic pelvic lymphoceles such as analgesics and/or lymphocele puncture and drainage.

3. Study Hypothesis We hypothesize that the intraoperative application of two collagen-fibrin patches (Tachosil®) to the obturator fossa and the femoral canal will reduce the number of symptomatic pelvic lymphoceles by at least 66% (primary study end point).

4. Study Design Prospective randomized clinical intervention trial of 140 women undergoing open or laparoscopic pelvic lymphadenectomy for cervical or endometrial cancer. Randomization will be by a computerized randomization list. Women will be centrally randomized by the principal investigator (CT). Allocation will be communicated by telephone after informed consent has been obtained and after lymphadenectomy has been completed. This is a single-blinded study, ie patients, but not surgeons, will be blinded to the treatment allocation. Outcome assessment will not be performed by the surgeon, who has performed the lymphadenectomy. Outcome assessors will be blinded to the treatment allocation.

5. Treatment

All women will undergo open or laparoscopic surgery. Within this procedure, as deemed appropriate by the surgeon, women will undergo pelvic lymphadenectomy. The procedure will be performed as follows:

The peritoneum will be incised parallel to the iliac vessels. Then, the iliac vessels will be screened for the presence of bulky lymph nodes. If a lymph node debulking is performed, no patch will be applied. In women who undergo routine pelvic lymphadenectomy, lymph node tissue will be removed from the external iliac vessels, the obturator fossa, the interiliac region, and the common iliac region after identification and appropriate preparation of surgical landmarks, ie iliac vessels, femoral canal, chorda, and obturator nerve. At the end of the procedure, hemostasis will be checked. A Tachosil® patch of 4.8x4.8cm will be attached to the obturator fossa and a Tachosil® patch of 4.8x4.8cm will be attached to the femoral canal of each side of surgery in the intervention group. In the control group, no Tachosil® patch will be used. No specific drainage of the retroperitoneum will be performed. All surgical procedures will be performed by the study team members Clemens Tempfer, Lukas Hefler, and Alexander Reinthaller, experienced in open and laparoscopic pelvic lymph node dissection. In order to ensure adequate application of the Tachosil® patch by laparoscopy, all surgeons will perform at least two laparoscopic training operations during which they roll the Tachosil® patch around a laparoscopic instrument, move it through a 10mm trocar into the abdomen, and flatten it out.

8. Statistical analysis A power calculation demonstrated that, with a sample size of 70 per group, a two-arm study has a power of 80% to detect a 66% absolute difference in treatment efficacy at a significance level of 0.05 regarding the primary outcome parameter, ie symptomatic lymphoceles CTCAE 4.03 grade >2. This calculation was based on published data by Tinelli et al. observing a rate of 32% of symptomatic lymphoceles in the placebo group and 10% in the Tachosil® group (5). Assuming a 10% drop out-rate, 140 women will be randomized. The chi-square test will used for comparisons of frequencies and cross-tabulations. One Way ANOVA on ranks will be used on means. Descriptive statistics (means, standard deviations, and ranges) will be used for demographic data. Bonferroni's correction will be used for multiple comparisons of secondary outcomes.

10. Follow-up All women will undergo a gynecologic examination and a transvaginal and transabdominal ultrasound examination at the time of discharge of the hospital, performed by a physician experienced in transvaginal and transabdominal ultrasound examinations, who has not participated in the original surgical procedure and is blinded to the treatment allocation. All women will be scheduled for a follow-up visit 4 weeks after surgery including a gynecologic examination and a transvaginal and transabdominal ultrasound examination, performed by a physician experienced in transvaginal and transabdominal ultrasound examinations, who has not participated in the original surgical procedure and is blinded to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing open or laparoscopic surgery for cervical or endometrial cancer
* Age between 18 and 70 yrs
* Informed consent

Exclusion Criteria:

* Women with previously diagnosed lymph edema
* Known disease of the lymphatic system
* Immunocompromised women such as those with an immunosuppressive medication or a known disease of the immune system

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
symptomatic lymph cysts | 4 weeks
  Primary outcome variable:
  2.1. To evaluate the incidence of symptomatic pelvic lymphoceles defined by CTCAE 4.03 grade >2 within 4 weeks after surgery in women undergoing open or laparoscopic pelvic lymphadenectomy for cervical and endometrial cancer with and without the application of Tachosil® during surgery.

SECONDARY OUTCOMES:
asymptomatic lymph cysts, intervention rate due to symptomatic lymph cysts | 4 weeks
  Secondary outcome variables:
  2.2. To evaluate the incidence of sonographically detected pelvic lymphoceles of at least 2cm in the largest diameter 4 weeks after surgery in women undergoing open or laparoscopic pelvic lymphadenectomy for cervical and endometrial cancer with and without the application of Tachosil® during surgery.
  2.3. To evaluate the rate and type of medical interventions for clinically symptomatic pelvic lymphoceles such as analgesics and/or lymphocele puncture and drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Tempfer, MD, Principal Investigator — Ruhr University Bochum, Germany
Locations (2):
- Medical University of Vienna, Vienna, Austria
- Ruhr University Bochum, Bochum, Germany

REFERENCES:
- [Background] O'Hanlan KA, Pinto RA, O'Holleran M. Total laparoscopic hysterectomy with and without lymph node dissection for uterine neoplasia. J Minim Invasive Gynecol. 2007 Jul-Aug;14(4):449-52. doi: 10.1016/j.jmig.2007.02.012. PMID 17630162
- [Background] Marchiole P, Benchaib M, Buenerd A, Lazlo E, Dargent D, Mathevet P. Oncological safety of laparoscopic-assisted vaginal radical trachelectomy (LARVT or Dargent's operation): a comparative study with laparoscopic-assisted vaginal radical hysterectomy (LARVH). Gynecol Oncol. 2007 Jul;106(1):132-41. doi: 10.1016/j.ygyno.2007.03.009. Epub 2007 May 9. PMID 17493666
- [Background] Xu H, Chen Y, Li Y, Zhang Q, Wang D, Liang Z. Complications of laparoscopic radical hysterectomy and lymphadenectomy for invasive cervical cancer: experience based on 317 procedures. Surg Endosc. 2007 Jun;21(6):960-4. doi: 10.1007/s00464-006-9129-0. Epub 2007 Feb 8. PMID 17287919
- [Background] Simonato A, Varca V, Esposito M, Venzano F, Carmignani G. The use of a surgical patch in the prevention of lymphoceles after extraperitoneal pelvic lymphadenectomy for prostate cancer: a randomized prospective pilot study. J Urol. 2009 Nov;182(5):2285-90. doi: 10.1016/j.juro.2009.07.033. Epub 2009 Sep 16. PMID 19762048
- [Background] Panici PB, Plotti F, Zullo MA, Muzii L, Manci N, Palaia I, Ruggiero A, Angioli R. Pelvic lymphadenectomy for cervical carcinoma: laparotomy extraperitoneal, transperitoneal or laparoscopic approach? A randomized study. Gynecol Oncol. 2006 Dec;103(3):859-64. doi: 10.1016/j.ygyno.2006.05.025. Epub 2006 Jun 27. PMID 16806442
- [Background] Frilling A, Stavrou GA, Mischinger HJ, de Hemptinne B, Rokkjaer M, Klempnauer J, Thorne A, Gloor B, Beckebaum S, Ghaffar MF, Broelsch CE. Effectiveness of a new carrier-bound fibrin sealant versus argon beamer as haemostatic agent during liver resection: a randomised prospective trial. Langenbecks Arch Surg. 2005 Apr;390(2):114-20. doi: 10.1007/s00423-005-0543-x. Epub 2005 Feb 19. PMID 15723234
- [Background] Anegg U, Lindenmann J, Matzi V, Smolle J, Maier A, Smolle-Juttner F. Efficiency of fleece-bound sealing (TachoSil) of air leaks in lung surgery: a prospective randomised trial. Eur J Cardiothorac Surg. 2007 Feb;31(2):198-202. doi: 10.1016/j.ejcts.2006.11.033. Epub 2006 Dec 21. PMID 17187983
- [Background] Siemer S, Lahme S, Altziebler S, Machtens S, Strohmaier W, Wechsel HW, Goebell P, Schmeller N, Oberneder R, Stolzenburg JU, Becker H, Luftenegger W, Tetens V, Van Poppel H. Efficacy and safety of TachoSil as haemostatic treatment versus standard suturing in kidney tumour resection: a randomised prospective study. Eur Urol. 2007 Oct;52(4):1156-63. doi: 10.1016/j.eururo.2007.04.027. Epub 2007 Apr 18. PMID 17467884
- [Background] Grimm C, Polterauer S, Helmy S, Cibula D, Zikan M, Reinthaller A, Tempfer C. A collagen-fibrin patch (Tachosil(R)) for the prevention of symptomatic lymphoceles after pelvic lymphadenectomy in women with gynecologic malignancies: a randomized clinical trial. BMC Cancer. 2014 Aug 30;14:635. doi: 10.1186/1471-2407-14-635. PMID 25175029
- [Result] Grimm C, Polterauer S, Helmy-Bader S, Zikan M, Cibula D, Heitz F, Harter P, Giese A, Reinthaller A, Tempfer C. A collagen-fibrin patch for the prevention of symptomatic lymphoceles after pelvic lymphadenectomy in women with gynecologic malignancies: A randomized clinical trial. Gynecol Oncol. 2018 Apr;149(1):140-145. doi: 10.1016/j.ygyno.2018.01.012. Epub 2018 Feb 12. PMID 29395308